CLINICAL TRIAL: NCT01944033
Title: β2-agonist Versus Ipratropium Bromide Associated With β2-agonists in Chronic Obstructive Pulmonary Disease Exacerbation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Pr. Semir Nouira, Semir Nouira, University of Monastir
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: β2-agonist
Record Dates: First submitted 2013-09-09; First posted 2013-09-17 (Estimated); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Acute Exacerbation of Chronic Obstructive Airways Disease
Keywords: β2-agonist; Ipratropium Bromide; Chronic Obstructive Pulmonary Disease Exacerbation; Emergency departement
MeSH Terms: interventions — Terbutaline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group Terbutaline (Active Comparator): Group Terbutaline received 5 mg Terbutaline sulfate (2ml) and 3ml serum saline in nebulization repeated three times during 1 hour and every 4 hours during the first 24 hour protocol
  Interventions: Drug: Bricanyl/Iprovent
- Group Terbutaline/IB (Experimental): Group Terbutaline/Ipratropium Bromide received combination of 5 mg Terbutaline (2ml) and 0.5 mg Ipratropium bromide (2ml) and 1ml serum saline in nebulization repeated threeand every 4 hours during the first 24 hour protocol
  Interventions: Drug: Bricanyl

INTERVENTIONS:
Drug: Bricanyl/Iprovent — 5 mg Terbutaline sulfate (2ml) + 0,5 mg Ipratropium bromide (2ml) + 1ml serum saline in each nebulization which is repeated three times during 1 hour and every 4 hours during the first 24 hour protocol
  Arms: Group Terbutaline
Drug: Bricanyl — 5 mg Terbutaline sulfate (2ml) + 3ml serum saline in each nebulization which is repeated three times during 1 hour and every 4 hours during the first 24 hour protocol
  Arms: Group Terbutaline/IB

SUMMARY:
The effectiveness of β2-agonists in the treatment of exacerbations of COPD is already established. The purpose of this study is to compare the effectiveness of the β2-agonists alone in nebulization with the association β2-agonists + Ipratropium bromide in the treatment of an acute exacerbation of COPD consulting the emergency departement based on the clinical and arterial blood gas.

DETAILED DESCRIPTION:
It is a prospective study and randomized performed in patients admitted to the emergency departement for acute exacerbation of COPD. The patients were divided in two groups: Group Terbutaline/Ipratropium Bromide; received Terbutaline + Ipratropium bromide in nebulization and Group Terbutaline received Terbutaline alone in nebulization)

ELIGIBILITY:
Inclusion Criteria:

* have known or suspected COPD based on pulmonary function test, arterial blood gas, clinical history, physical examination, and chest radiograph
* Age over 18 years old.
* COPD Exacerbation: sustained worsening of patient's condition from stable state necessitating change in regular medication within the last two weeks and need for non invasive ventilation with regard to arterialo blood gas abnormalities: PaCO2 > 45 mmHg, PH<7,35 SaO2<90%

Exclusion Criteria:

* GCS ≤ 14
* hypersensitivity to anticholinergic
* severe acidosis
* immediate need for intubation
* lack of patient cooperation
* serious hemodynamic unstability or systolic blood pressure < 90 mmHg, heart arrhythmia

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2013-07; Primary Completion 2016-07 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
hospital admission rate and ICU admission rate | within 24 hours after ED admission

SECONDARY OUTCOMES:
dyspnea score | 24 hours after ED admission
endotracheal intubation rate | within 24 hours after ED admission

CONTACTS AND LOCATIONS:
Overall Officials: semir nouira, Pr, Principal Investigator — University of Monastir
Locations (2):
- Tunisia (2):
  - University Hospital of Monastir, Monastir, Monastir Governorate
  - Fattouma Bourguiba University Hospital, Monastir

IPD SHARING:
Plan to Share IPD: Yes